CLINICAL TRIAL: NCT05566717
Title: An Investigator-Initiated Study to Assess the Association of Diabetic Retinopathy Severity Scale (DRSS) With Level of Decreased Corneal Sensitivity
Acronym: Assess
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Center Ophthalmology Associates (Other)
Collaborators: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASSESS
Record Dates: First submitted 2022-08-02; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Diabetic Retinopathy; Neurotrophic Keratitis
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the association between level of decreased corneal sensitivity and diabetic retinopathy severity scale

DETAILED DESCRIPTION:
This study is assessing the association between neurotrophic keratopathy and diabetic retinopathy severity by examining subjects with diabetic retinopathy to associate DRSS and disease characteristics with corneal desensitization. In addition, to better understand the relationship of disease duration, HbA1c, and status of concurrent systemic therapies and diabetic retinopathy treatments, predictive modelling will be performed to determine predictive factors of patients at highest risk of developing reduced corneal sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 1 or Type 2 diabetes with DRSS of 3 or higher
* Be willing and able to sign the informed consent form (ICF)
* Be at least 18 years of age
* Be literate and able to complete questionnaires independently
* Have provided verbal and written informed consent

Exclusion Criteria:

* Have a history of vitrectomy
* Have a history of cornea, eyelid, glaucoma, or retina surgery
* Have a history of previously diagnosed neurotrophic keratopathy or other cranial nerve V pathology, such as trigeminal neuralgia
* Have a history of ocular herpes simplex virus infection
* Have a history of herpes zoster ophthalmicus
* Have a history of ocular chemical trauma
* Have a history of underlying corneal dystrophies
* Have had cataract surgery less than 3 months prior
* Have a history of pan-retinal photocoagulation (PRP)
* Have current Stage 2 or 3 neurotrophic keratopathy
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to Visit 1

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a single-center, controlled study to assess the association of diabetic retinopathy severity with reduction in corneal sensitivity in approximately 50 Type 1 and Type 2 diabetes subjects (100 eyes) at least 18 years of age and meeting all other study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 3months
  • To associate the Diabetic Retinopathy Severity Scale level 3 or higher (as confirmed by masked reading center) with the level of decreased corneal sensitivity in patients with Type 1 and Type 2 diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center Ophthalmology Associates, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared however demographics and baseline characteristics will be summarized.